CLINICAL TRIAL: NCT05125926
Title: Safety, Reactogenicity, and Immunogenicity of a SARS-CoV-2 Vaccine LYB001 in Healthy Adults: a Randomized, Double Blinded, Placebo-controlled Phase Ⅰ Trial
Brief Title: A Phase Ⅰ Trial to Evaluate the Safety and Immunogenicity of SARS-CoV-2 Vaccine LYB001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB001/CT-LAO-101
Record Dates: First submitted 2021-11-12; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- low-dose LYB001 in participants aged 18-59 years (Experimental): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: LYB001
- Placebo comparator Ⅰ in participants aged 18-59 years (Placebo Comparator): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: Placebo
- high-dose LYB001 in participants aged 18-59 years (Experimental): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: LYB001
- Placebo comparator Ⅱ in participants aged 18-59 years (Placebo Comparator): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: Placebo
- low-dose LYB001 in participants aged over 60 years (Experimental): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: LYB001
- Placebo comparator Ⅲ in participants aged over 60 years (Placebo Comparator): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: Placebo
- high-dose LYB001 in participants aged over 60 years (Experimental): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: LYB001
- Placebo comparator Ⅳ in participants aged over 60 years (Placebo Comparator): Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LYB001 — The investigational vaccine, with its antigen consisting of receptor-binding domain (RBD) from SARS-CoV-2 and virus-like particle (VLP) vector, adjuvanted with aluminum hydroxide. The investigational are administered through Intramuscular injection (IM) at upper arm deltoid on day 0, 28, 56.
  Arms: high-dose LYB001 in participants aged 18-59 years; high-dose LYB001 in participants aged over 60 years; low-dose LYB001 in participants aged 18-59 years; low-dose LYB001 in participants aged over 60 years
Biological: Placebo — Aluminum hydroxide
  Arms: Placebo comparator Ⅰ in participants aged 18-59 years; Placebo comparator Ⅱ in participants aged 18-59 years; Placebo comparator Ⅲ in participants aged over 60 years; Placebo comparator Ⅳ in participants aged over 60 years

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase Ⅰ trial in healthy adults aged 18 years and older, intended to evaluate the safety, reactogenicity, and immunogenicity profile of LYB001. The study vaccine will be administered IM at upper arm deltoid as a three-dose regimen with 28d interval on day 0, 28, 56.

To ensure the safety of the participants, the phase Ⅰ trial was will be carried out in a dose-escalation and age-sequential enrolment manner:

1. The safety, reactogenicity, and immunogenicity will be firstly evaluated in a cohort of adults aged 18-59 years randomly assigned (4:1) either to receive low-dose (25µg) LYB001 or placebo. After confirmation of an favorable 7-day safety, reactogenicity profile in this cohort by investigator, the study was able to proceed to the cohort of adults aged 18-59 years receiving high-dose (50µg) LYB001 or placebo.
2. After completing a favorable 7-day safety observation following the first dose of 50μg LYB001 in cohorts aged 18-59 years, the study was able to advance to cohorts aged ≥ 60 years receiving low-dose (25µg) LYB001 or placebo.

By analogy, all dose and age-stratified groups will be sequentially enrolled. The study will be ended after all participants completed 360-day safety observation following the 3rd dose of vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 years and older;
2. Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
3. For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).
4. Body mass index within range of 18~30 kg/m2.

Exclusion Criteria:

1. Abnormal results of laboratory screening tests which was clinically significant judged by clinicians;
2. Abnormal vital signs with clinical significance at screening, with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, or axillary body temperature ≥ 37.3°C;
3. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
4. History of human coronavirus infection/diseases, such as severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
5. History of COVID-19, or history of close contact with confirmed/suspected COVID-19 patients, or positive results for either SARS-CoV-2 nucleic acid or antibody tests (IgG and IgM) at screening;
6. Administration of antipyretics or painkillers within 24 hours prior to vaccination;
7. Receipt of any COVID-19 vaccine, live attenuated vaccine within 28 days prior to vaccination and other vaccines, such as subunit and inactived vaccine within 14 days prior to vaccination;
8. Receipt of blood or blood-related products, including immunoglobulins, within 3 months prior to vaccination; or any planned use during the study period.
9. Subjects with the following diseases:

   1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
   2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
   3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
   4. Currently suffering from or previously diagnosed with infectious diseases, positive screening results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus antibody；
   5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
   6. Asplenia, or functional asplenia；
   7. Presence of severe, uncontrollable or hospitalization indicated cardiovascular diseases, diabetes, neurological diseases (e.g., Guillain-Barre syndrome), blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
   8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
10. Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
11. History of a major surgery, per the investigator's judgment, within 12 weeks before vaccination, or not achieving full recovery after surgery, or any planned major surgery during the study;
12. Pregnant or lactating females, or those who plan to become pregnant during the study period;
13. Having participated or being participating in COVID-19 related clinical trials, and those being participating or planning to participate in other clinical trials during the study period;
14. Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 28 days after each dose
  Immediate adverse events (AEs) within 30 minutes after each vaccination, solicited local and systemic AEs for within 7 days and unsolicited AEs within 28 days following each vaccination;1. Immediate adverse events (AEs) within 30 minutes after each vaccination, solicited local and systemic AEs for within 7 days and unsolicited AEs within 28 days following each vaccination;

SECONDARY OUTCOMES:
Serious adverse events (SAEs) | 360 days after first vaccination
  Serious adverse events (SAEs) throughout the study
Safety laboratory measures | 3 days after each dose
  Changes of safety laboratory measures and vital signs at day 3 following each vaccination in comparison to pre-vaccination levels.
Geometric neutralizing titers (GMT), Geometric Mean Increases (GMI) and seroconversion rates against wild-type SARS-CoV-2 | pre dose 1, day 14 post dose 2, day 14, 28 post dose 3
  Geometric neutralizing titers (GMT), Geometric Mean Increases (GMI) and seroconversion rates against wild-type SARS-CoV-2
GMT, GMI and seroconversion rates against SARS-CoV-2 variants of concern (VOCs) | pre dose 1, day 14 post dose 2, day 14, 28 post dose 3
  GMT, GMI and seroconversion rates against SARS-CoV-2 variants of concern (VOCs)
GMT, GMI and seroconversion rates of S protein-binding antibodies | pre dose 1, day 14 post dose 2, day 14, 28 post dose 3
  GMT, GMI and seroconversion rates of S protein-binding antibodies
Cellular Immune Response | pre dose 1, day 14 post dose 2, day 14 dose 3
  1. Th1 and Th2 immune responses by enzyme-linked immunospot (ELISPOT) assay, Th1: interferon gamma (IFN-γ), interleukin-2 (IL-2), Th2: IL-4, IL-6.

IPD SHARING:
Plan to Share IPD: No